CLINICAL TRIAL: NCT01900704
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter Study to Investigate the Efficacy and Safety of SER120 Nasal Spray Formulation in Patients With Nocturia
Brief Title: Multicenter Study to Investigate SER120 Nasal Spray Formulations in Patients With Nocturia - DB4
Acronym: DB4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serenity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPC-SER120-DB4-201301
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2015-11

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SER120 750 ng (Experimental): SER120 750 ng
  Interventions: Drug: SER120 750 ng
- SER120 1500 ng (Experimental): SER120 1500 ng
  Interventions: Drug: SER120 1500 ng
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SER120 750 ng — SER120 750 ng
  Arms: SER120 750 ng
Drug: SER120 1500 ng — SER120 1500 ng
  Arms: SER120 1500 ng
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To investigate the efficacy and safety of SER120 nasal spray formulations in patients with nocturia

ELIGIBILITY:
Inclusion Criteria:

* Male and female 50 years or older
* Nocturia of 6 or more months duration averaging greater than 2 nocturic episodes per night

Exclusion Criteria:

* CHF
* Diabetis Insipidus
* Renal insufficiency
* Hepatic insufficiency
* Incontinence
* Illnesses requiring systemic steroids
* Malignancy within the past 5 years
* Sleep apnea
* Nephrotic syndrome
* Unexplained pelvic mass
* Urinary bladder neurological dysfunction
* Urinary bladder surgery or radiotherapy
* Pregnant or breast feeding

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stephen M. Auerbach, MD, Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SER120 1500 ng: All participants received SER120 1500 ng once daily
- SER120 750 ng: All participant received SER120 750 ng once daily
- Placebo: All participants received Placebo once daily
Period: Overall Study
Arm/Group | SER120 1500 ng | SER120 750 ng | Placebo
Started | 270 | 270 | 270
Completed | 229 | 235 | 237
Not Completed | 41 | 35 | 33

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat Population
Groups:
- SER120 750 ng: All participants received SER120 750 ng once daily
- Total: Total of all reporting groups
Arm/Group | SER120 750 ng | SER120 1500 ng | Placebo | Total
Number analyzed (Participants) | 262 | 260 | 260 | 782
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (8.8) | 66.1 (9.2) | 65.8 (9.0) | 66.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 113 | 114 | 344
  Male | 145 | 147 | 146 | 438
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 6 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 26 | 40 | 39 | 105
  White | 229 | 212 | 220 | 661
  More than one race | 3 | 2 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 247 | 238 | 249 | 734
  Canada | 15 | 22 | 11 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Nocturic Episodes at the End of Treatment Compare to Prior to Treatment
Description: Change was calculated based on the number of mean nocturic episodes per night between baseline through week 12
Time Frame: 12 weeks
Population: intent to treat population
Measure: Least Squares Mean (Standard Error); unit: nocturic episodes per night
Arm/Group | SER120 750 ng | SER120 1500 ng | Placebo
Number analyzed (Participants) | 262 | 260 | 260
nocturic episodes per night | -1.4 (0.06) | -1.5 (0.06) | -1.2 (0.06)

2. Primary Outcome: Percent of Participants With Equal of Greater Than 50% Reduction in Mean Nocturic Episodes
Description: Percent of participants with equal of greater than 50% reduction in mean nocturic episodes over the twelve week period
Time Frame: 12 weeks
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Groups:
- SER120 1500 ng: All participant received SER120 1500 ng once daily
Arm/Group | SER120 750 ng | SER120 1500 ng | Placebo
Number analyzed (Participants) | 262 | 260 | 260
Participants | 93 | 121 | 74

ADVERSE EVENTS:
Description: Adverse events were collected from the Safety Population, i.e., any patient who had received one dose of study drug and reported an adverse event.
Arm/Group | SER120 750 ng | SER120 1500 ng | Placebo
Serious Adverse Events (participants affected / at risk) | 7/266 | 4/264 | 5/267
Other Adverse Events (participants affected / at risk) | 30/266 | 30/264 | 30/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 750 ng (N=266) | SER120 1500 ng (N=264) | Placebo (N=267)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gallbladder empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 750 ng (N=266) | SER120 1500 ng (N=264) | Placebo (N=267)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 14 (14) | 18 (18)
Urinary tract infection (Infections and infestations) | 12 (12) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 8 (8) | 11 (11) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes